CLINICAL TRIAL: NCT03968796
Title: TENS and Kinesio Tape for Treatment Lateral Epicondylitis
Brief Title: Efficacy of Transcutaneous Electrical Nerve Stimulation (TENS) and Kinesio Taping in Patients With Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Lefke (Other)
Responsible Party: Principal Investigator, Hilal Telli, Assistant Professor - Medical Doctor, European University of Lefke
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Lateral Epicondylitis
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Pain in Arm, Unspecified; Tenosynovitis Elbow; Lateral Epicondylitis (Tennis Elbow) Bilateral
Keywords: Kinesio Taping; Lateral epicondylitis; Tennis elbow; TENS
MeSH Terms: conditions — Tennis Elbow | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator): A total of 10 sessions of TENS were administered to each patient for 20 minutes daily.
  Kinesio taping was performed a total of 3 sessions on the 1st, 4th and 7th days of treatment.
  Interventions: Other: Transcutaneous Electrical Nerve Stimulation (TENS); Other: Kinesio Taping
- Group 2 (Active Comparator): A total of 10 sessions of TENS were administered to each patient for 20 minutes daily.
  Sham Kinesio taping was performed a total of 3 sessions on the 1st, 4th and 7th days of treatment, but taping was done incorrectly.
  Interventions: Other: Transcutaneous Electrical Nerve Stimulation (TENS); Other: Sham Kinesio Taping
- Group 3 (Active Comparator): A total of 10 sessions of Sham TENS(the device was not operated) were administered to each patient for 20 minutes daily.
  Kinesio taping was performed a total of 3 sessions on the 1st, 4th and 7th days of treatment.
  Interventions: Other: Sham Transcutaneous Electrical Nerve Stimulation (TENS); Other: Kinesio Taping
- Group 4 (Placebo Comparator): A total of 10 sessions of Sham TENS(the device was not operated) were administered to each patient for 20 minutes daily.
  Sham Kinesio taping was performed a total of 3 sessions on the 1st, 4th and 7th days of treatment, but taping was done incorrectly.
  Interventions: Other: Sham Transcutaneous Electrical Nerve Stimulation (TENS); Other: Sham Kinesio Taping

INTERVENTIONS:
Other: Transcutaneous Electrical Nerve Stimulation (TENS)
  Arms: Group 1; Group 2
Other: Sham Transcutaneous Electrical Nerve Stimulation (TENS)
  Arms: Group 3; Group 4
Other: Kinesio Taping
  Arms: Group 1; Group 3
Other: Sham Kinesio Taping
  Arms: Group 2; Group 4

SUMMARY:
Lateral epicondylitis is the most common condition affecting the elbow and characterized by pain over the lateral epicondyle. The aim of this study was to determine and compare the efficacy of TENS and Kinesio Taping in lateral epicondylitis.

DETAILED DESCRIPTION:
In this prospective-randomized, assessor blinded controlled trial, seventy-eight patients (63 women, 15 men, mean age 47,5 ±7,94 years) with lateral epicondylitis were enrolled. Patients were allocated into 4 treatment groups: Group 1 received TENS and Kinesio Taping, group 2 received TENS+sham Kinesio Taping, group 3 received sham TENS+ Kinesio Taping and group 4 received sham TENS+sham Kinesio Taping. TENS was applied for 10 sessions and Kinesio Taping for 4 times in 10 days. All patients were given a progressive exercise program and were informed about the disease. All patients were told to take paracetamol 500 mg if their pain is severe and to note the number of the paracetamol taken.

Outcome measures were pain-free grip strength, pressure pain threshold and pain severity at rest, night and forced wrist extension test. Patient-rated tennis elbow evaluation (PRTEE) was used to determine functional status. Patients were assessed for outcome measures at screening, after treatment (day 10) and 12th week after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19 to 72
* Enough cognitive ability to fill clinical assessment forms
* Agreed to participate in the study

Exclusion Criteria:

* Severe or progressive neurological deficits
* Severe psychiatric disease history, substance and/or alcohol dependence,
* Uncontrolled diabetes mellitus, malignancy, osteoporosis
* A history of inflammatory or infectious disease
* A skin allergy story
* Previously undergone physical therapy due to lateral epicondylitis

Ages: 19 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2013-08-31 (Actual); Study Completion 2013-08-31 (Actual)

PRIMARY OUTCOMES:
Pain-free grip strength | 12 week
  Hand grasping force with hand dynamometer was evaluated. The grip force was measured with the hand dynamometer as the maximum grip force, while the patient was sitting in the chair with 0 degrees of abduction and neutral position and the elbow with 90 degrees of flexion. Both sides were firstly measured on 2 sides and then averaged. 30 second rest periods were given between measurements.Patients were assessed for outcome measures at screening, after treatment (day 10) and 12th week after the treatment.
Pain severity at rest, night and forced wrist extension test | 12 week
  Pain was evaluated with a 10 cm scale horizantal VAS. The head of the line was painless and the end was the most severe pain. The patient was asked to mark the most appropriate location for pain on the scale. Pain severity at rest, at night and forced wrist extension test was evaluated by visual analog scale (VAS). Patients were assessed for outcome measures at screening, after treatment (day 10) and 12th week after the treatment.
Pressure pain threshold | 12 week
  Pressure pain threshold was evaluated by algometer. The pressure pain threshold was measured at the lateral epicondyle with an algae before starting with a painless side in both extremities. Algometer is an instrument that measures the pain threshold and pain tolerance objectively. In the sitting position, the shoulder is evaluated at 30 ° abduction, and the elbow at 90 ° flexion over the lateral epicondyle (1 cm 2 area).
  In our study, the algometer was applied vertically to the most painful point by increasing the pressure by 1 kg / cm2 every 3 seconds until the patient felt pain. The pressure value that caused the pain feeling was determined as the pain threshold. In the 20-second intervals, the lowest pressure value was taken as the pain threshold between the three measurements. Patients were assessed for outcome measures at screening, after treatment (day 10) and 12th week after the treatment.
Patient-rated tennis elbow evaluation (PRTEE) | 12 week
  Patient-rated tennis elbow evaluation (PRTEE)was used to determine functional status. The PRTEE (Patient Based Inventory Evaluation Questionnaire) is a practical questionnaire that measures elbow pain and function and has been validated in lateral epicondylitis. It consists of a total of 15 questions about pain, function and daily activities. In our study, pain, function and total score were calculated for each patient. The pain score is obtained by summing the points given to the 5 questions related to the pain in the affected arm (minimum score 0, maximum score 50). Function score is obtained by dividing the scores of 10 questions evaluating the function in the affected arm and dividing by 2 (minimum score 0, maximum score 50). The total score is the sum of the pain score and function score (minimum score 0, maximum score of 100).Patients were assessed for outcome measures at screening, after treatment (day 10) and 12th week after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Telli, MD, Principal Investigator — European University of Lefke

IPD SHARING:
Plan to Share IPD: No
Patients were allocated into 4 treatment groups: Group 1 received TENS and Kinesio Taping, group 2 received TENS + sham Kinesio Taping, group 3 received sham TENS + Kinesio Taping and group 4 received sham TENS + sham Kinesio Taping. TENS was applied for 10 sessions and Kinesio Taping for 4 times in 10 days. All patients were given a progressive exercise program and were informed about the disease. All patients were told to take paracetamol 500 mg if their pain is severe and to note the number of the paracetamol taken. Outcome measures were pain-free grip strength, pressure pain threshold and pain severity at rest, night and forced wrist extension test. Patient-rated tennis elbow evaluation (PRTEE) was used to determine functional status. Patients were assessed for outcome measures at screening, after treatment (day 10) and 12th week after the treatment.